CLINICAL TRIAL: NCT06716788
Title: Development and Clinical Translation of Protein-losing Enteropathy (PLE) Imaging PET Probe
Brief Title: 68Ga-HSA PET/CT Imaging for Protein-losing Enteropathy
Acronym: PLE-PET
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Suzhou Transcenta Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: 2023YJZ61
Record Dates: First submitted 2024-01-15; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-12

CONDITIONS: Cancer
Keywords: PET/CT; Protein-Losing Enteropathy; 68Ga labeling; Human serum albumin
MeSH Terms: conditions — Neoplasms; Protein-Losing Enteropathies

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- 68Ga-HSA PET/CT in participants with hypoproteinemia: Participants who are with hypoproteinemia will be injected with 2.22 MBq/kg body weight of 68Ga-HSA in one dose intravenously and then undergo PET/CT scan within 1 h.
  Interventions: Drug: 68Ga-HSA

INTERVENTIONS:
Drug: 68Ga-HSA — 68Ga-HSA PET/CT: after intravenous injection of 2.22 MBq/kg body weight of quality-controlled 68Ga-HSA, a Siemens Biograph PET/CT scan will be applied within 1 h, and the scan range will be from the top of the head to 1/3 of the upper thigh.
  Other Names: 68Ga-DTPA-HSA

SUMMARY:
In this project, based on the DTPA-HAS kit, investigators plan to develop a positron nuclide 68Ga labeled DTPA-HSA molecular probe in order to obtain high sensitivity, signal-to-noise ratio and high-resolution PET/CT imaging images, aiming to find the specific site of intestinal leakage while diagnosing Protein-Losing Enteropathy (PLE), and analyze the pathological mechanism of intestinal leakage in combination with pathology, so as to provide molecular imaging guidance for the treatment of PLE patients. PLE is a rare gastrointestinal protein-losing syndrome, and the radiopharmaceutical 99mTc-DTPA-HSA (99mTc-human serum albumin) approved by the State Food and Drug Administration has the diagnostic ability of protein-losing enteropathy (PLE), but due to the low resolution of SPECT/CT, the image clarity and signal-to-noise ratio need to be improved, it is a classic probe in the last century, unable to meet the existing clinical needs.

DETAILED DESCRIPTION:
This project developed a a new type of nuclide Ga-68 labeled DTPA-HSA probe, and with the inherent advantages of this nuclear medicine department, it has promoted the formulation of the production filing standard of the drug, and obtained the 68Ga-HSA injection that can be used for preclinical research and meets the clinical standards. Clinical research on 68Ga-HSA PET/CT imaging was carried out to provide a basis for the diagnosis and treatment of PLE patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with digestive system tumors;
2. Presence of hypoproteinemia or clinical manifestations of hypoplasma protein;
3. Serum albumin <30 g/L, AAT>80 ml/d;
4. Measurable lesions in imaging;
5. Predicted survival greater than 3 months;

Exclusion Criteria:

1. Severe hepatic or renal dysfunction;
2. Pregnant or nursing;
3. Known allergy to the investigational drug or its excipients in study;
4. Unable to comply with the PET/CT imaging procedures;
5. Claustrophobia or other psychiatric disorders;
6. Other conditions deemed unsuitable for participation in the trial;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients at Being Cancer Hospital who are confirmed protein-losing enteropathy, or digestive system tumors with hypoproteinemia.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Standard Uptake Value Value | 1 year
  The standardized uptake value(SUV) of 68Ga-HSA in suspected PLE lesions measured by the PET/CT
SUVR | 1 year
  Ratio of the SUV of 68GA-DTPA-HSA in the suspected PLE lesions to the SUV of 68Ga DTPA-HSA in the normal tissues corresponding to the PLE (SUVR)

CONTACTS AND LOCATIONS:
Overall Officials: Hua Zhu, Study Director — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No